CLINICAL TRIAL: NCT05601687
Title: Endoscopic Step-up Approach Vs Aggressive Debridement of Large Pancreatic Walled-off Necrosis - a Single-center, Open-label, Randomized, Superiority Trial (ACCELERATE)
Brief Title: Endoscopic Step-up Approach Vs Aggressive Debridement of Large Pancreatic Walled-off Necrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Gitte Aabye Olsen, MD, Principle Investigator, MD, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Accelerate
Record Dates: First submitted 2022-10-21; First posted 2022-11-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Necrosis; Pancreatitis, Acute Necrotizing
Keywords: Walled-off necrosis; Walled-off pancreatic necrosis; Endoscopic necrosectomy; Video-assisted retroperitoneal debridement
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Intervention Model Description: Patients shall be randomly assigned in a 1:1 ratio to either the step-up or the accelerated approach. Block randomization shall be performed with a concealed, fixed block size using a web-based randomization program. Random block sizes of 4 or 6 shall be used for preparation of the randomization sequence. The computer-generated block randomization assignments shall be placed in opaque sealed envelopes. Randomization shall be performed by a study coordinator when patients meet the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step-up Approach (Active Comparator): Standard procedure where necrosectomy is only performed in the absence of clinical improvement 72 hours after placements of lumen-apposing metal stent.
  Interventions: Procedure: Step-up Approach
- Direct Endoscopic Necrosectomy (Experimental): Necrosectomy will be performed in the same procedure as the placement of the lumen-apposing metal stent.
  Interventions: Procedure: Direct Endoscopic Necrosectomy

INTERVENTIONS:
Procedure: Direct Endoscopic Necrosectomy — Endosonography-guided, transmural drainage of the WONs shall be performed using a lumen-apposing metal stent (LAMS).After placement of the LAMS, EN shall be performed during the same procedure (Direct EN). After DEN, a 7-Fr/4cm double pigtail and a 7-Fr nasocystic irrigation catheter shall be placed through the LAMS. Endoscopic necrosectomy and VARD shall be repeated as often as clinically indicated and logistically possible with a minimum of one day between procedures
  Arms: Direct Endoscopic Necrosectomy
Procedure: Step-up Approach — Endosonography-guided, transmural drainage of the WONs shall be performed using a lumen-apposing metal stent (LAMS). After placement of the LAMS, a 7-Fr/4cm double pigtail stent and a 7-Fr nasocystic catheter shall be placed through the LAMS.
  The effect of the index drainage procedure shall be evaluated every 72 hours and next treatment step will depend on whether the patient's condition improves.
  If clinical improvement is observed, the drainage regime continues, and no further therapeutic action shall be taken.
  In absence of clinical improvement after 72 hours and if supplementary drainage is impossible, the patient shall proceed to endoscopic necrosectomy (EN) or video-assisted retroperitoneal debridement (VARD). Absence of clinical improvement due to causes not related to the WON treatment, e.g., urinary tract or pulmonary infection or iv catheter sepsis, shall not influence the treatment algorithm of the WON.
  Arms: Step-up Approach

SUMMARY:
The goal of this clinical trial is to compare a conventional endoscopic step-up approach with an accelerated treatment algorithm using direct endoscopic necrosectomy in patients with acute necrotizing pancreatitis and walled of necroses exceeding a diameter of 15 cm. It will be investigated whether an aggressive treatment algorithm instead of a classical step-up approach will shorten the length of stay in the hospital and also reduce the mortality in patients treated for large walled off necroses.

DETAILED DESCRIPTION:
INTRODUCTION While most patients with acute pancreatitis suffer a mild and uncomplicated course of disease, up to 20% develop a more severe course with development of pancreatic and/or peripancreatic necroses. With time, these necroses become encapsulated with a well-defined inflammatory wall, so called walled-off necroses (WONs). Up to 30% of WONs become infected, which prolongs the length of hospital stay (LOS), increases morbidity and mortality significantly, and generally requires some kind of invasive intervention. During the last two decades, a minimally invasive step-up approach consisting of percutaneous and/or endoscopic, transluminal drainage followed, if necessary, by percutaneous, video-assisted retroperitoneal debridement (VARD) or endoscopic necrosectomy (EN), have replaced open surgery as the standard treatment resulting in improved patient outcomes. Copenhagen University Hospital Hvidovre have for nearly two decades treated more than 400 WON patients with an actual annual number of 40-50 patients. This center serves as a tertiary referral center, the only in East-Denmark, with a background population of 2.6 million. In line with international guidelines, endoscopic step-up approach has been practiced as standard care for infected WONs. This approach follows international recommendations of delaying index procedures until at least four weeks after debut of pancreatitis (to ensure encapsulation) and then only applying the least invasive intervention needed. The decision to step-up is triggered by absence of biochemical and/or clinical improvement or clinical deterioration.

Recently, lumen-apposing metal stents (LAMS) have been introduced for the transluminal treatment of pancreatic fluid collections. The stent is fully-covered and shaped with two bilateral anchor flanges with a saddle in between. A dedicated through-the-scope delivery system, where the tip serves as an electrocautery device enables extra-luminal access and deployment of the stent. Conventionally, transmural drainage with installation of two double pigtail plastic stents (DPS) has been the method of choice. Although drainage with plastic stents seems non-inferior to LAMS, the DPS method implies a need for repetitive dilatation of the drainage tract because of spontaneous closure of the tract and thereby probably a higher number of endoscopic procedures. By keeping the transmural tract patent, LAMS may improve drainage and facilitate endoscopic necrosectomy, which may even be performed during the index procedure (direct endoscopic necrosectomy (DEN)).

The LOS is considerable for patients treated for infected WON, especially those with complex and large fluid collections. Copenhagen University Hvidovre Hospital has one of the largest prospective single center databases registering all patients treated with WON. The median LOS for patients with large WONs exceeding 15 cm in diameter treated with the step-up approach, is 58 days. During the hospital stay, patients undergo weekly endoscopic or surgical procedures, and many patients additionally need treatment in the intensive care unit. Together, the treatment of patients with WON carries a substantial economic burden for the health care system. Furthermore, even in a tertiary care setting, the mortality is still up to 15% in complex cases with large fluid collections. The mortality in patient needing treatment in intensive care unit (ICU) is much higher, nearly 40%. Unprotocolized cases with urgent needs for an augmented course of treatment (e.g. cases with malignancy demanding surgery or oncological therapy) have been successfully treated with an accelerated treatment algorithm. Likewise, an international multicenter study found that an aggressive treatment was safe with promising results. The invastegators hypothesize, that a general alteration in the treatment algorithm instigating an aggressive treatment algorithm instead of a classical step-up approach might not only shorten LOS, but also reduce the mortality in patients treated for large WONs.

AIM To compare a conventional endoscopic step-up approach with an accelerated treatment algorithm using DEN.

STUDY DESIGN A single-center open-label, randomized, controlled 2 armed superiority study.

Patients with acute, necrotizing pancreatitis and WON exceeding a diameter of 15 cm will be randomized to either the endoscopic step-up approach or direct endoscopic necrosectomy.

The primary endpoint is a composite of death, major complications occurring within 6 months following randomization, or length of stay exceeding 58 days.

From results previously published by Copenhagen University Hospital Hvidovre, it is shown that the risk of death for eligible patients is estimated to 5%, the risk of major complications is 5%, while the risk of exceeding a LOS of above 58 days is 50%. The investigators assume that the risk of death and major complications will remain at 5% and 5%, respectively, while the rate of patients exceeding a LOS of 58 days will be reduced by 75% to 12.5%. Based on these estimates, 48 patients are required to have an 80% change (5% significant level) of detecting an increase in success rate in the primary outcome measure from 40% in the control group to 77.5% in the interventional group.

The investigators will after inclusion of 25 patients conduct an interim analysis to assess whether one of the study groups are superior to an extent that will ethically call for an early termination of the study. Likewise, safety will continually be assessed in conjunction with the ethics committee.

ELIGIBILITY:
Inclusion Criteria:

All criteria must be fulfilled

1. Patients with acute, necrotizing pancreatitis and

   * WON exceeding a diameter of 15 cm.
   * Imaging test(s) must be done within 1 week before the index drainage procedure.
   * Debut of pancreatitis must be within 3 months before the index drainage procedure.
2. One or more indication(s) for endoscopic, transmural drainage must be established:

   1. Confirmed or suspected infection.
   2. Severe intraabdominal hypertension or abdominal compartment syndrome.
   3. Persisting abdominal pain, early satiety, or general discomfort.
   4. Obstruction of the GI or biliary tract.
   5. Leakage of pancreatic juice, e.g. pancreatic ascites or pleural effusion.
3. Preoperatively, the WON must be considered eligible for endoscopic, transgastric drainage. Distance between the gastric wall and WON must not exceed one cm and there must be no major interposed vessels.

Exclusion Criteria:

1. Patients under the age of 18.
2. Pregnancy.
3. Known or suspected malignant disease.
4. Pancreatitis secondary to trauma or surgical intervention.
5. Chronic pancreatitis.
6. Previous surgical or endoscopic drainage or necrosectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
A composite of major complications, death, or length of stay exceeding 58 days | From date of randomization until discharge, assessed up to 12 months
  If patients either die, encounter a major complication, or stay in hospital for longer than 58 days, it will be registered as an event.
  Major complications are defined as new onset (i.e. not present 24 hours before randomization) organ failure (cardiovascular, pulmonary or renal), bleeding requiring intervention, perforation of a visceral organ requiring intervention, enterocutaneous fistula requiring intervention and incisional hernia (including burst abdomen).

SECONDARY OUTCOMES:
Length of hospital stay from the index drainage procedure | From date of randomization until discharge, assessed up to 12 months
Total number of debridement procedures | From date of randomization until discharge, assessed up to 12 months
  Number of endoscopic necrosectomies and video-assisted retroperitoneal debridements needed throughout the disease course.
Total number of endoscopic procedures | From date of randomization until discharge, assessed up to 12 months
Total number of drainage and debridement procedures (radiological, endoscopic, and surgical) | From date of randomization until discharge, assessed up to 12 months
Number of days from index drainage procedure until removal of naso-cystic catheter | From date of randomization until discharge, assessed up to 12 months
Duration of drainage and debridement procedures (index and cumulated) measured in minutes | From date of randomization until discharge, assessed up to 12 months
Days at the hospital during a 6-month follow up | Assessed up to 12 months following randomization
Length of ICU stay | From date of randomization until discharge, assessed up to 12 months
  Days in the ICU during hospitalization
Number of days until resolution of pre-interventional systemic inflammatory response syndrome (SIRS) | From date of randomization until discharge, assessed up to 12 months
  Number of days from randomization to restoration of normal blood pressure, temperature, heart rate, inspiratory rate, and white blood cell count
New onset episodes of culture verified bacteremia | From date of randomization until discharge, assessed up to 12 months
Occurrence of splanchnic vein thrombosis (portal-, splenic-, or superior mesenteric vein) | From date of randomization until discharge, assessed up to 12 months
  Portal-, splenic-, or superior mesenteric vein thrombosis
Need for tube feeding (naso-gastric or naso-jejunal) or parenteral nutrition | From date of randomization until discharge, assessed up to 12 months
CRP-area under curve | From date of randomization until discharge, assessed up to 12 months
  AUC from the index drainage procedure until discharge from hospital
Number of adverse events | From date of randomization until discharge, assessed up to 12 months
  according to the ASGE lexicon and Clavien-Dindo
Mortality | From date of randomization until discharge, assessed up to 12 months
  The rate mortality compared between the two study groups
Unset of exocrine and endocrine insufficiency | From date of randomization until discharge, assessed up to 12 months
  The unset of diabetes and/or steatorrhea
Total treatment costs. | From date of randomization until discharge, assessed up to 12 months
  In euros and dollars

CONTACTS AND LOCATIONS:
Overall Officials: John G Karstensen, MD Ph.d., Study Director — Pancreatitis Centre East (PACE), Gastro Unit, Copenhagen University Hospital Hvidovre, Denmark
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Sharing upon reasonable request
Supporting Information: Study Protocol
Access Criteria: Sharing upon reasonable request

REFERENCES:
- [Background] Ebrahim M, Werge MP, Hadi A, Lahchich M, Nagras ZG, Lauritsen ML, Schmidt PN, Hansen EF, Novovic S, Karstensen JG. Clinical outcomes following endoscopic or video-assisted retroperitoneal management of acute pancreatitis with large (>15 cm) walled-off pancreatic necrosis: Retrospective, single tertiary center cohort study. Dig Endosc. 2022 Sep;34(6):1245-1252. doi: 10.1111/den.14295. Epub 2022 Mar 29. PMID 35258123
- [Background] Banks PA, Freeman ML; Practice Parameters Committee of the American College of Gastroenterology. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006 Oct;101(10):2379-400. doi: 10.1111/j.1572-0241.2006.00856.x. No abstract available. PMID 17032204
- [Background] van Brunschot S, van Grinsven J, Voermans RP, Bakker OJ, Besselink MG, Boermeester MA, Bollen TL, Bosscha K, Bouwense SA, Bruno MJ, Cappendijk VC, Consten EC, Dejong CH, Dijkgraaf MG, van Eijck CH, Erkelens GW, van Goor H, Hadithi M, Haveman JW, Hofker SH, Jansen JJ, Lameris JS, van Lienden KP, Manusama ER, Meijssen MA, Mulder CJ, Nieuwenhuis VB, Poley JW, de Ridder RJ, Rosman C, Schaapherder AF, Scheepers JJ, Schoon EJ, Seerden T, Spanier BW, Straathof JW, Timmer R, Venneman NG, Vleggaar FP, Witteman BJ, Gooszen HG, van Santvoort HC, Fockens P; Dutch Pancreatitis Study Group. Transluminal endoscopic step-up approach versus minimally invasive surgical step-up approach in patients with infected necrotising pancreatitis (TENSION trial): design and rationale of a randomised controlled multicenter trial [ISRCTN09186711]. BMC Gastroenterol. 2013 Nov 25;13:161. doi: 10.1186/1471-230X-13-161. PMID 24274589
- [Background] Seewald S, Groth S, Omar S, Imazu H, Seitz U, de Weerth A, Soetikno R, Zhong Y, Sriram PV, Ponnudurai R, Sikka S, Thonke F, Soehendra N. Aggressive endoscopic therapy for pancreatic necrosis and pancreatic abscess: a new safe and effective treatment algorithm (videos). Gastrointest Endosc. 2005 Jul;62(1):92-100. doi: 10.1016/s0016-5107(05)00541-9. PMID 15990825
- [Derived] Olsen GA, Schmidt PN, Hadi A, Prahm AP, Werge MP, Roug S, Schefte DF, Lauritsen ML, Hansen EF, Novovic S, Karstensen JG. Accelerated vs Step-Up Endoscopic Treatment for Pancreatic Walled-Off Necrosis: A Randomized Controlled Trial (ACCELERATE). Clin Gastroenterol Hepatol. 2025 Aug 18:S1542-3565(25)00701-3. doi: 10.1016/j.cgh.2025.08.007. Online ahead of print. PMID 40835042
- See also: Related Info — https://www.hvidovrehospital.dk/Research/pace/Pages/default.aspx